CLINICAL TRIAL: NCT02366988
Title: Phase 3 Prospective, Multicentric Randomized Study of Endoscopic Versus Surgical Treatment of Bile Duct Stricture in Chronic Pancreatitis
Brief Title: The PASTEC Study: Endoscopic Stenting Versus Surgery for the Treatment of Bile Duct Stricture in Chronic Pancreatitis
Acronym: PASTEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decision: not enough inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012_43; 2013-A01671-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-09-24; First posted 2015-02-20 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic pancreatitis; Clinical Trial; Bile stricture; Endoscopy; Surgery
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic Biliary Stenting (Active Comparator): Temporary self-expandable metallic covered stent
  Interventions: Device: Endoscopic Biliary Stenting
- Surgical treatment (Active Comparator): Bilio-enteric anastomosis including Whipple, Frey or Beger procedure, double or triple derivation
  Interventions: Procedure: Surgical treatment Bilio-enteric anastomosis

INTERVENTIONS:
Device: Endoscopic Biliary Stenting — Endoscopic probe self-expandable metallic covered stent Biliary stent will be left in place for 6 months
  Arms: Endoscopic Biliary Stenting
Procedure: Surgical treatment Bilio-enteric anastomosis — Bilio-enteric anastomosis including Whipple, Frey or Beger procedure, double or triple derivation
  Arms: Surgical treatment

SUMMARY:
Biliary obstruction complicates the course of chronic pancreatitis in 3%-23% of patients and in these cases, endoscopy and surgery are the treatment modalities of choice. Morbid-mortality of these procedures is similar and physicians face the decision between endoscopy and surgery for this group of patients, with no randomized controlled trial available comparing these procedures.

The PASTEC trial is a multicenter, phase III, randomized, comparing the effectiveness of surgical and endoscopic interventions in the management of bile duct stricture for chronic pancreatitis.

The primary end point is 18-months normalization of serum alkaline phosphatase. Secondary end points are morbid-mortality rate, quality of life, numbers of endoscopic or surgical procedures, length of stay. Eighty-six patients need to be included.

DETAILED DESCRIPTION:
This study is planned to last for 4 years, with a 2-year inclusion period and a 2-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptomatic chronic pancreatitis-related biliary duct stricture (pain or jaundice or pale stool / dark urine)
* Biological symptomatic chronic pancreatitis-related biliary duct stricture (elevation of serum alkaline phosphatase (>2 or 3 times the upper limit of normal values) and/or of serum bilirubin for longer than 1 month)
* Isolated biliary stricture or biliary stricture associated to main pancreatic duct stricture
* Secondary biliary cirrhosis
* Progression of biliary stricture

Exclusion Criteria:

* Pancreatic malignancy
* Cirrhosis
* Portal vein thrombosis, portal cavernoma
* Primary sclerosing cholangitis
* Recent acute pancreatitis (i.e., in the previous 3 weeks)
* Acute hepatitis
* Post-surgical biliary stricture
* Biliary stones or pseudocyst-related biliary duct stricture
* Previous pancreatic surgery or endoscopic sphincterotomy
* Score IV or V on the American Society of Anesthesiologists scale
* Pregnancy or breastfeeding
* Patient aged under 18 yrs
* Emergency clinical situations (i.e., angiocholitis with septicemia)
* Non-compliant patients or suffering from legal incapacity
* Contra-indication for endoscopic or surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
normalization of serum alkaline phosphatase (considered as < 130 UI/L) | 18 months
  A normal value of serum alkaline phosphatase will be considered as < 130 UI/L

SECONDARY OUTCOMES:
Quality of Life (EORTC health surveys) | At 18 months
  EORTC health surveys will administered to assess quality of life.
abdominal pain (Clinical symptoms assessed by Izbicki's score) | at 1, 3, 6, 12,18 months after the procedure
  Clinical symptoms assessed by Izbicki's score,
jaundice, (Clinical symptoms assessed) | at 1, 3, 6, 12,18 months after the procedure
  Clinical symptoms assessed
pruritus, (Clinical symptoms assessed) | at 1, 3, 6, 12,18 months after the procedure
  Clinical symptoms assessed
pale stool, (Clinical symptoms assessed) | at 1, 3, 6, 12,18 months after the procedure
  Clinical symptoms assessed
dark urine. (Clinical symptoms assessed) | at 1, 3, 6, 12,18 months after the procedure
  Clinical symptoms assessed
Cholestasis | At 1, 3, 6, 12, 18 months after the procedure
  Biological measures Cholestasis Bilirubinemia < 1,2 mg/dl (norms : 0,1 à 1,2 mg / dl) Gamma GT < 50 UI / L
Cytolysis | At 1, 3, 6, 12, 18 months after the procedure
  Biological measures Cytolysis TGO < 40 UI / L (norms : 15 à 40 UI / L) TGP < 40 UI / L (norms : 10 à 40 UI / L)
Liver failure | At 1, 3, 6, 12, 18 months after the procedure
  Biological measures Liver failure TP > 60% (norms : 60 à 120%) Facteur V > 60% (norms : 60 à 120%)
CT-Scan (Morphological assessment) | At 6 and 18 months after the procedure
  Morphological assessment by CT-Scan, Pseudocyst, main pancreatic duct > 3 mm, inflammatory cephalic mass > 4 cm, biliary duct stricture, pancreatic calcifications
Bili-MRI | At 6 and 18 months after the procedure
  Morphological assessment by Bili-MRI, Pseudocyst, main pancreatic duct > 3 mm, inflammatory cephalic mass > 4 cm, biliary duct stricture, pancreatic calcifications
presence of surgical complications ( dindo and Clavien ) | At 1, 3, 6, 12, 18 months
Hospital length of stay | At 1, 3, 6, 12, 18 months
number of re - hospitalization | At 1, 3, 6, 12, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ZERBIB, MD, PhD, Study Chair — University Hospital, Lille
Locations (7):
- France (7):
  - Centre hospitalier, Béthune
  - Centre hospitalier, Dunkirk
  - Centre Hospitalier Dr Schaffner, Lens
  - Clinique de la Louvière, Lille
  - Hôpital St Philibert, Lomme
  - Centre hospitalier, Roubaix
  - Centre hospitalier, Valencienne